CLINICAL TRIAL: NCT00752895
Title: A Randomized, Double-Blind, Placebo Controlled Trial of North American Ginseng Extract (CVT-E002; COLD-fX®) to Prevent Respiratory Infection and Reduce Antibiotic Use in Patients With Chronic Lymphocytic Leukemia
Brief Title: American Ginseng Extract in Preventing Respiratory Infection and in Reducing Antibiotic Use in Patients With CLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00006819; U10CA081851 (NIH); REBACCCWFU98308 (Other: NCI)
Record Dates: First submitted 2008-09-13; First posted 2008-09-16 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I - Ginseng (Experimental): Patients receive oral American ginseng extract twice daily.
  Interventions: Dietary Supplement: American ginseng
- Arm II - Placebo (Placebo Comparator): Patients receive oral placebo twice daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: American ginseng — Given orally
  Arms: Arm I - Ginseng
Dietary Supplement: Placebo — Given orally
  Arms: Arm II - Placebo

SUMMARY:
RATIONALE: American ginseng extract may prevent or reduce acute respiratory illness in patients with chronic lymphocytic leukemia. It is not yet known whether American ginseng extract is more effective than a placebo in preventing respiratory infections.

PURPOSE: This randomized trial is studying the side effects of American ginseng extract and to see how well it works compared with a placebo in preventing respiratory infection and in reducing antibiotic use in patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effect of American ginseng extract on the number of days of acute respiratory infection (ARI) during the peak respiratory illness season (January-March) in patients with chronic lymphocytic leukemia (CLL).
* To determine the safety of American ginseng extract in these patients evaluated according to NCI CTCAE v3.0.

Secondary

* To assess the effect of this treatment on antibiotic use days (AUDs).
* To assess the effect of this treatment on the rate of all infections diagnosed by a physician.
* To assess the effect of this treatment on the duration and severity of each ARI episode.
* To assess the effect of this treatment on major infections defined as infection severe enough to require hospitalization or intravenous antibiotics.
* To assess the effect of this treatment on the incidence of herpes zoster infection defined as an episode of physician-diagnosed zoster infection.
* To assess the effect of this treatment on CLL disease activity (i.e., serum IgG, total lymphocyte count, platelet count, and Rai staging).
* To determine the incidence of ARI and type of illness in an untreated cohort of CLL patients over an entire winter respiratory illness season (January 1- April 30).

Tertiary

* To determine the effect of this treatment on the incidence of influenza and respiratory syncytial virus confirmed by a physician.

OUTLINE: This is a multicenter study. Patients are stratified according to antibiotic prophylaxis with trimethoprim-sulfamethoxazole (yes vs no), serum IgG (≤ 500 mg/dL vs > 500 mg/dL), and influenza vaccine status (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral American ginseng extract twice daily.
* Arm II: Patients receive oral placebo twice daily. Treatment in both arms continues for up to 4 months in the absence of illness or adverse events.

After completion of study treatment, patients are followed at 4 weeks by phone.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL)

  * Phenotypic evidence (i.e., flow cytometry or bone marrow biopsy) of disease
* Untreated CLL allowed

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 months
* Creatinine < 2.0 mg/dL OR creatinine clearance > 50 mL/min
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception prior to and during study treatment
* No known cirrhosis, collagen vascular disease, multiple sclerosis, or HIV positivity
* No other prior or concurrent malignancies except for non-melanoma skin cancers or carcinoma in situ of the cervix

  * Other prior malignancies allowed provided the patient has been disease-free for > 5 years
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No psychiatric or social illness that would limit compliance with study requirements
* No history of allergy or other adverse response to ginseng products
* No history of seasonal or environmental allergies that require ongoing treatment with antihistamines, intranasal corticosteroids, or systemic corticosteroids

PRIOR CONCURRENT THERAPY:

* More than 3 months since prior and no concurrent chlorambucil
* At least 1 month since prior and no other concurrent herbal ginseng products
* No prior or concurrent fludarabine, alemtuzumab, rituximab, intravenous immunoglobulin, or hematopoietic stem cell transplantation
* No concurrent corticosteroids (20 mg/day of prednisone or equivalent)
* No concurrent antibiotic prophylaxis, except for trimethoprim-sulfamethoxazole
* No concurrent warfarin
* No other concurrent investigational or commercial agents or other therapies with the intent to treat the patient's malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2009-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin High, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (125):
- United States (125):
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - St. Vincent Oncology Center, Indianapolis, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I - Ginseng | Arm II - Placebo
Started | 147 | 146
Completed | 139 | 143
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 8 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Ginseng | Arm II - Placebo | Total
Number analyzed (Participants) | 147 | 146 | 293
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 64 | 135
  >=65 years | 76 | 82 | 158
Age, Continuous [Median (Full Range); unit: years] | 65 [43 to 87] | 66 [44 to 82] | 65 [43 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 60 | 125
  Male | 82 | 86 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 147 | 144 | 291
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 145 | 141 | 286
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 147 | 146 | 293

OUTCOME MEASURES:

1. Primary Outcome: Acute Respiratory Infection (ARI) Days
Description: An ARI day was defined as any day for which the subject experienced one or more respiratory symptoms (cough, sore throat, nasal or sinus congestion, or runny nose) and one or more systemic symptoms (feverishness, chills/sweats, myalgia (muscle aches), fatigue, headache, poor endurance or increased shortness of breath) between January and March.
Time Frame: 3 months
Population: Participants who returned a respiratory symptom diary between January and March. Note that a few participants failed to provide respiratory diaries so the numbers of participants for these analyses do not necessarily match the numbers who remained in the study or the numbers with adverse event data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I - Ginseng | Arm II - Placebo
Number analyzed (Participants) | 137 | 143
days | 8.30 (16.87) | 6.78 (13.27)
Statistical Analysis 1: Comparison: Arm I - Ginseng vs Arm II - Placebo; Test type: Superiority or Other; p = 0.295, Negative binomial regression — This p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05

2. Secondary Outcome: Number of Antibiotic Use Days
Description: An antibiotic day was defined as a day on which the subject took one or more antibiotics between January and March.
Time Frame: 3 months
Population: Participants who returned respiratory symptom and antibiotic use diaries. Note that a few participants failed to provide antibiotic use diaries so the numbers of participants for these analyses do not necessarily match the numbers who remained in the study or the numbers with adverse event data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I - Ginseng | Arm II - Placebo
Number analyzed (Participants) | 137 | 143
days | 1.12 (3.42) | 1.55 (6.46)
Statistical Analysis 1: Comparison: Arm I - Ginseng vs Arm II - Placebo; Test type: Superiority or Other; p = 0.820, Negative binomial regression — This p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05

ADVERSE EVENTS:
Time Frame: 5 months
Description: Note that some participants had adverse events and later dropped out so the numbers of participants for these analyses do not necessarily match the numbers who remained in the study or the numbers with primary outcome data.
Arm/Group | Arm I - Ginseng | Arm II - Placebo
Serious Adverse Events (participants affected / at risk) | 11/140 | 16/143
Other Adverse Events (participants affected / at risk) | 121/140 | 126/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Ginseng (N=140) | Arm II - Placebo (N=143)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cardiac ischemia/fnfarction (Cardiac disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea - without colostomy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage, GI: Peritoneal cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (2) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Infection with Grade 3/4 ANC: Skin (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or grade 1/2 neutrophils: Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1/2 neutrophils: Spleen (Infections and infestations) | 0 (0) | 1 (2)
Infection with unknown ANC: upper airway NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC: Brain (encephalitis) (Infections and infestations) | 1 (1) | 0 (0)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (5)
Pain: Abdomen NOS (General disorders) | 0 (0) | 3 (4)
Pain: Back (General disorders) | 0 (0) | 1 (1)
Pain: Chest Wall (General disorders) | 0 (0) | 2 (2)
Pain: Chest/thorax NOS (General disorders) | 0 (0) | 1 (1)
Pain:Stomach (General disorders) | 0 (0) | 1 (1)
Platelets (160-360) (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Pleural Effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Cardiac disorders) | 1 (1) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary Frequency / Urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Frequency / Urgency - Pllakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Ventricular Arrhythmia NOS (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Ginseng (N=140) | Arm II - Placebo (N=143)
Diarrhea - without colostomy (Gastrointestinal disorders) | 15 (22) | 19 (25)
Dizziness (Nervous system disorders) | 17 (27) | 18 (24)
Hyperglycemia (Metabolism and nutrition disorders) | 32 (56) | 44 (70)
Headache (Nervous system disorders) | 38 (58) | 39 (63)
Heartburn (Gastrointestinal disorders) | 27 (46) | 36 (57)
Hemorrhage, Nose - Epistaxis (General disorders) | 3 (4) | 11 (15)
Hypertension (Cardiac disorders) | 21 (34) | 23 (37)
Insomnia (Psychiatric disorders) | 55 (85) | 36 (63)
Nausea (Gastrointestinal disorders) | 8 (9) | 14 (18)
Neurology - Other - Nervousness (Nervous system disorders) | 18 (22) | 11 (15)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 57 (110) | 65 (123)
Rash / Desquamation (Skin and subcutaneous tissue disorders) | 6 (6) | 13 (20)
Urinary Frequency / Urgency - Pllakiuria (Renal and urinary disorders) | 40 (77) | 33 (54)
Vomiting (Gastrointestinal disorders) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes